CLINICAL TRIAL: NCT06344988
Title: The Effect of Online Exercise Program on Musculoskeletal Problems, Upper Extremity Function, Physical Activity Level, Muscle Oxygenation, Reaction Time, Grip Strength and Pressure Pain Threshold in Musicians Playing Stringed Instruments
Brief Title: Physical and Functional Effects of Online Exercise Program on Musicians Playing Stringed Instruments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Sule Kecelioglu, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/41-10
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Diseases or Conditions; Musculoskeletal Pain
Keywords: musicians playing stringed instruments
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A 40-minute online education presentation will be given on the role of postural and dynamic muscles, the importance of physical activity, the gradual adaptation of the body to workload and physical stressors, rest, and injury management. They will also be asked to wear a smart band. Additionally, the exercise program developed by Chan et al., will be practised online via "Google Meet" once a week for 8 weeks, each session lasting 40-45 minutes.
  Interventions: Other: The exercise program; Other: Online education presentation; Device: Smart band
- Control Group (Other): A 40-minute online education presentation will be given on the role of postural and dynamic muscles, the importance of physical activity, the gradual adaptation of the body to workload and physical stressors, rest, and injury management. They will also be asked to wear a smart band.
  Interventions: Other: Online education presentation; Device: Smart band

INTERVENTIONS:
Other: The exercise program — The exercise program developed by Chan et al., consists of a 30-minute exercise period with 5 minute warm-up (diaphragmatic breathing, general body movements) and 5-10 minute cool-down (stretching exercises in addition to the exercises in the warm-up period) periods. Exercises include 6 steps and 5 series (neck, shoulder, spine, abdominals, hip) according to difficulty level. The total exercise program takes 40-45 minutes.
  Arms: Intervention Group
Other: Online education presentation — This online education presentation includes the role of postural and dynamic muscles, the importance of physical activity, gradual adaptation of the body to workload and physical stressors, rest, and injury management. The education takes 40 minutes and will be done once.
Device: Smart band — Participants will be given a Xiaomi Mi Smart Band 5 and will be asked not to remove the smart band except for bathing for 8 weeks, and to download the smart phone application (Zepp Life) compatible with the smart band to their phones, which will allow their steps to be recorded on a weekly basis.

SUMMARY:
Musculoskeletal problems related to instrument playing or performance are frequently seen in musicians. Different interventions such as strength training, endurance training and yoga have been used in the management of these problems. The first specific exercise program for professional orchestra musicians was developed by Chan et al. However, it has been stated that it is difficult to encourage musicians' participation in exercise due to their constantly changing work schedules, and at this point, the use of digital media such as DVDs, USBs, and educational exercise videos may have a potential role.

On the other hand, it has been stated that smart wearable devices with mobile applications (such as smart watches, smart band) as digital health interventions are an interesting, interactive and efficient psychological strategy to promote physical activity and can be used as an intervention to promote a healthy lifestyle. Based on the literature, in our study, the exercise program developed by Chan et al., will be done online via "Google Meet" and symptoms can be evaluated with objective evaluation methods. Unlike other studies using digital media, exercises will be performed synchronously and feedback will be given to the musicians simultaneously, as in face-to-face exercises. In addition, all participants will be given a smart band, they will be encouraged to use it until the end of the study, and the change in their physical activity levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Agreeing to exercise once a week for 8 weeks
* Being between the ages of 18-65
* Playing a string instrument in Bursa Regional State Symphony Orchestra / Bursa Uludağ University State Conservatory / Bursa Uludağ University Faculty of Education Fine Arts Education Department, Department of Music Education / Ege University State Conservatory of Turkish Music
* Main instrument being a stringed instrument (violin, viola, cello, double bass)
* Playing an instrument for more than 5 years
* Having a musculoskeletal problem related to playing an instrument or performance

Exclusion Criteria:

* Having a musculoskeletal problem that is not related to playing an instrument or performance
* Playing the instrument less than 15 hours per week
* Having had a corticosteroid injection within 6 weeks
* Having used anti-inflammatory or gabapentin within 3 weeks
* Having had any surgical operation that would prevent exercise in the last 6 months
* Having any diagnosed neurological and/or orthopedic problem that would prevent exercise in the last 6 months
* Having a diagnosed psychiatric problem
* Maximum subcutaneous fat thickness more than 12 mm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal problems | baseline and 8 weeks after baseline
  The Cornell Musculoskeletal Discomfort Questionnaire will be used to evaluate musculoskeletal problems. The questionnaire includes visuals of different parts of the body, and in these parts, the frequency and severity of pain, ache or discomfort felt by the person within a week, and whether it prevents work are questioned separately. The Turkish validity of the questionnaire was found to be good at .62-.92, and the test-retest reliability was found to be adequate at .56-.97. A high score from the questionnaire indicates that musculoskeletal problems are intense.
Muscle oxygenation | baseline and 8 weeks after baseline
  The Moxy muscle oxygen monitor is a lightweight and small device that measures regional blood flow and oxygenation by placing it on the skin non-invasively using near infrared spectroscopy (NIRS). The Moxy muscle oxygen monitor has been shown to be a valid and reliable device in terms of muscle oxygenation compared to other NIRS devices. Its validity in measuring muscle oxygenation (SROC: r = 0.842-0.993, ICC: r = 0.773-0.992, p < .01) was found to be strong or very good, and its reliability was moderate to high in low-intensity exercise. The left deltoid muscle will be evaluated in musicians. The evaluation will be made at rest (3 minutes), in the instrument holding position (3 minutes), during the instrument playing position (3 minutes) and at rest after playing the instrument (3 minutes).
  Note: The maximum subcutaneous fat thickness that the device can measure is 12 mm. A skinfold caliper will be used to identify participants who will be excluded from the study.
Pressure pain threshold | baseline and 8 weeks after baseline
  Pressure pain threshold, defined as the minimum force that triggers pain, is measured with a tool called an algometer. The value obtained when the person indicates the time when the feeling of pressure turns into a painful feeling is recorded in kg/cm2. The lower the value, the lower the person's pressure pain threshold. In the reliability study of the algometer device, the ICC value was found to be high at = 0.91. For musicians, evaluations will be taken from the right and left trapezius muscle and the right and left lateral epicondyle.
Reaction time | baseline and 8 weeks after baseline
  BlazePod™ will be used to measure reaction time. It was stated that the ICC value was 0.82. A lighting protocol is created via the mobile application for the use of the device. In this device, which consists of sensors, the time taken for the participants to turn off the visual stimulus is recorded in milliseconds. The device planned to be used in the study will consist of 3 sensors. There will be 2 simple and 1 choice reaction time assessments. For simple reaction time, the participants' right hand will be evaluated first, then their left hand (with a blue light on the sensor). For choice reaction time, participants will be asked to use their right hand when the blue light is on and their left hand when the red light is on. Participant reaction time data will be accessed via the BlazePod mobile application.
Grip strength | baseline and 8 weeks after baseline
  Saehan dynamometer will be used to measure grip strength. The evaluation will be made with the elbow in 90° flexion and the forearm in a neutral position, which is the standard test position of the American Association of Hand Therapists. Evaluations will be made in 3 repetitions on the right and left hands and the average of the obtained values will be taken. Test-retest reliability was found to be excellent for the Saehan dynamometer (r=0.981 right hand and r=0.985 left hand).

SECONDARY OUTCOMES:
Upper extremity function | baseline and 8 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) will be used to evaluate upper extremity function. The Turkish validity and reliability study of the DASH was conducted by Düger et al. A high score from the DASH results indicates a high level of disability.
Physical activity level | baseline and 8 weeks after baseline
  Physical activity level will be evaluated both with the data obtained from the smart band and the International Physical Activity Questionnaire Short Form (IPAQ-SF).
  Smart band: Participants' weekly step count will be recorded with Xiaomi Mi Smart Band 5. They will be asked to download the smart phone application (Zepp Life) for iOS or Android, which is compatible with the smart band to phones.
  International Physical Activity Questionnaire Short Form (IPAQ-SF): The Turkish validity and reliability study of the questionnaire was conducted by Saglam et al. The questionnaire evaluates the time spent on vigorous and moderate physical activity, walking and sitting in the last 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Selnur Narin Aral, Assoc. Prof., Study Director — Dokuz Eylul University
Locations (4):
- Turkey (Türkiye) (4):
  - Bursa Regional State Symphony Orchestra, Bursa
  - Bursa Uludağ University Faculty of Education Fine Arts Education Department, Department of Music Education, Bursa
  - Bursa Uludağ University State Conservatory, Bursa
  - Ege University State Conservatory of Turkish Music, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan C, Driscoll T, Ackermann B. Development of a specific exercise programme for professional orchestral musicians. Inj Prev. 2013 Aug;19(4):257-63. doi: 10.1136/injuryprev-2012-040608. Epub 2012 Dec 4. PMID 23211353
- [Background] Chan C, Driscoll T, Ackermann B. Exercise DVD effect on musculoskeletal disorders in professional orchestral musicians. Occup Med (Lond). 2014 Jan;64(1):23-30. doi: 10.1093/occmed/kqt117. Epub 2013 Nov 9. PMID 24213243
- [Background] Roos M, Roy JS. Effect of a rehabilitation program on performance-related musculoskeletal disorders in student and professional orchestral musicians: a randomized controlled trial. Clin Rehabil. 2018 Dec;32(12):1656-1665. doi: 10.1177/0269215518785000. Epub 2018 Jun 29. PMID 29954190
- [Background] Yen HY. Smart wearable devices as a psychological intervention for healthy lifestyle and quality of life: a randomized controlled trial. Qual Life Res. 2021 Mar;30(3):791-802. doi: 10.1007/s11136-020-02680-6. Epub 2020 Oct 26. PMID 33104939
- [Background] Zaza C, Charles C, Muszynski A. The meaning of playing-related musculoskeletal disorders to classical musicians. Soc Sci Med. 1998 Dec;47(12):2013-23. doi: 10.1016/s0277-9536(98)00307-4. PMID 10075243
- [Background] Erdinc O, Hot K, Ozkaya M. Turkish version of the Cornell Musculoskeletal Discomfort Questionnaire: cross-cultural adaptation and validation. Work. 2011;39(3):251-60. doi: 10.3233/WOR-2011-1173. PMID 21709361
- [Background] Jester A, Harth A, Wind G, Germann G, Sauerbier M. Disabilities of the arm, shoulder and hand (DASH) questionnaire: Determining functional activity profiles in patients with upper extremity disorders. J Hand Surg Br. 2005 Feb;30(1):23-8. doi: 10.1016/j.jhsb.2004.08.008. PMID 15620487
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Crum EM, O'Connor WJ, Van Loo L, Valckx M, Stannard SR. Validity and reliability of the Moxy oxygen monitor during incremental cycling exercise. Eur J Sport Sci. 2017 Sep;17(8):1037-1043. doi: 10.1080/17461391.2017.1330899. Epub 2017 May 30. PMID 28557670
- [Background] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Background] de-Oliveira LA, Matos MV, Fernandes IGS, Nascimento DA, da Silva-Grigoletto ME. Test-Retest Reliability of a Visual-Cognitive Technology (BlazePod) to Measure Response Time. J Sports Sci Med. 2021 Mar 1;20(1):179-180. doi: 10.52082/jssm.2021.179. eCollection 2021 Mar. No abstract available. PMID 33708001